CLINICAL TRIAL: NCT04558450
Title: Covid-19 Effects on ARTErial StIffness and Vascular AgiNg
Brief Title: Covid-19 Effects on Arterial Stiffness and Vascular Aging (CARTESIAN)
Acronym: CARTESIAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: The Association for Research into Arterial Structure and Physiology (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200762; APHP200762 (Other: ANSM); 20.07.24.57438 (Other: CNRIPH)
Record Dates: First submitted 2020-08-31; First posted 2020-09-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Covid19; Arterial Stiffness; Endothelial Dysfunction; Diastolic Dysfunction
MeSH Terms: conditions — COVID-19 | interventions — Carotid-Femoral Pulse Wave Velocity

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Other): Patients with confirmed infection by SARS-Cov-2, requiring a hospitalization in intensive care unit
  Interventions: Diagnostic Test: carotid-femoral pulse-wave velocity
- Group 2 (Other): Patients with confirmed infection by SARS-Cov-2, requiring a hospitalization in a medicine unit
  Interventions: Diagnostic Test: carotid-femoral pulse-wave velocity
- Group 3 (Other): Patients with confirmed infection by SARS-Cov-2, not requiring hospitalization
  Interventions: Diagnostic Test: carotid-femoral pulse-wave velocity
- Group 4 (Other): 4) individuals having performed a test for SARS-Cov-2 infection, but resulted to be negative
  Interventions: Diagnostic Test: carotid-femoral pulse-wave velocity

INTERVENTIONS:
Diagnostic Test: carotid-femoral pulse-wave velocity — early vascular aging tests
  Other Names: arterial distensibility; wave separation/intensity analysis; flow-mediated dilation; cardiac diastolic dysfunction; myocardial stiffness; central blood pressure

SUMMARY:
The purpose of the study is to evaluate the presence of early vascular aging 6 months and 12 months after COVID-19 infection.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all eligible patients giving written informed consent will undergo a comprehensive non-invasive assessment of vascular and cardiac function 6 months and 12 months after COVID-19 infection. Cardiovascular events and mortality will be collected 2, 5 and 10 years after inclusion

ELIGIBILITY:
Inclusion Criteria:

* age >18 years, both sexes;
* written informed consent;
* affiliation to a social security regime;
* a recent diagnosis of COVID19 (6±3 months) proven by PCR or serology (for group 1,2,3)
* hospitalization in intensive care unit for COVID19 (for group 1)
* hospitalization in a medicine unit for COVID19 (for group 2)
* no hospitalization for COVID19 or hospitalization less than 24h (for group 3)
* a negative test for SARS-nCOV2 infection (PCR or serology)(for group 4)

Exclusion Criteria:

* Age <18 years
* Inability to express consent of the study
* Diseases carrying out a life -expectancy <1 year according to clinical judgment
* Pregnancy and breastfeeding
* Foreseen inability to attend scheduled visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
PWV | 6 months after COVID19 infection
  carotid-femoral pulse wave velocity measured by application tonometry
PWV | 12 months after COVID19 infection
  carotid-femoral pulse wave velocity measured by application tonometry
PWV change | difference between PWV at 12 and 6 months after COVID19 infection
  carotid-femoral pulse wave velocity measured by application tonometry

SECONDARY OUTCOMES:
arterial distensibility | 6 months after COVID19 infection
  carotid, radial and digital distensibility by standard and ultrahigh frequency ultrasound
arterial distensibility | 12 months after COVID19 infection
  carotid, radial and digital distensibility by standard and ultrahigh frequency ultrasound
arterial distensibility change | difference between arterial distensibility at 12 and 6 months after COVID19 infection
  carotid, radial and digital distensibility by standard and ultrahigh frequency ultrasound
brachial artery FMD | 6 months after COVID19 infection
  brachial artery flow-mediated dilation for non-invasive evaluation of endothelial dysfunction, by ultrasound and automatic edge detection analysis
brachial artery FMD | 12 months after COVID19 infection
  brachial artery flow-mediated dilation for non-invasive evaluation of endothelial dysfunction, by ultrasound and automatic edge detection analysis
brachial artery FMD change | difference between FMD at 12 and 6 months after COVID19 infection
  brachial artery flow-mediated dilation for non-invasive evaluation of endothelial dysfunction, by ultrasound and automatic edge detection analysis
central blood pressure | 6 months after COVID19 infection
  central blood pressure obtained non-invasively by application tonometry and validated transfer function
central blood pressure | 12 months after COVID19 infection
  central blood pressure obtained non-invasively by application tonometry and validated transfer function
central blood pressure (BP) change | difference between central BP at 12 and 6 months after COVID19 infection
  central blood pressure obtained non-invasively by application tonometry and validated transfer function
wave separation/wave intensity analysis (WSA/WIA) | 6 months after COVID19 infection
  peripheral arterial waveform analysis aimed at exploring wave reflection and micro-macrocirculation crosstalk
wave separation/wave intensity analysis (WSA/WIA) | 12 months after COVID19 infection
  peripheral arterial waveform analysis aimed at exploring wave reflection and micro-macrocirculation crosstalk
WSA/WIA change | difference between WSA/WIA at 12 and 6 months after COVID19 infection
  peripheral arterial waveform analysis aimed at exploring wave reflection and micro-macrocirculation crosstalk
cardiac diastolic dysfunction | 6 months after COVID19 infection
  E/e' at rest and after low-level exercise
cardiac diastolic dysfunction | 12 months after COVID19 infection
  E/e' at rest and after low-level exercise
cardiac diastolic dysfunction change | difference between cardiac diastolic dysfunction at 12 and 6 months after COVID19 infection
  E/e' at rest and after low-level exercise
myocardial stiffness | 6 months after COVID19 infection
  cardioelastography by ultrafast ultrasound
myocardial stiffness | 12 months after COVID19 infection
  cardioelastography by ultrafast ultrasound
myocardial stiffness change | difference between myocardial stiffness at 12 and 6 months after COVID19 infection
  cardioelastography by ultrafast ultrasound
carotid femoral and hearth carotid change | 6 months after COVID19 infection
  Mesure by laser doppler vibrometry

OTHER OUTCOMES:
total mortality | 2 years
  individual data will be meta-analyzed with sister studies running in parallel worldwide
total mortality | 5 years
  individual data will be meta-analyzed with sister studies running in parallel worldwide
total mortality | 10 years
  individual data will be meta-analyzed with sister studies running in parallel worldwide
CV events | 2 years
  fatal+non-fatal
CV events | 5 years
  fatal+non-fatal
CV events | 10 years
  fatal+non-fatal

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUTOUYRIE, MD PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - CHRU Nancy, Nancy
  - Hôpital Européen Georges Pompidou - APHP, Paris
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.

REFERENCES:
- See also: general description of the study — http://www.arterysociety.org/our-activities-2/cartesian-2/
- See also: summary and presentation of the global CARTESIAN initiative — http://vascagenet.eu/successful-information-session-on-the-cartesian-study